CLINICAL TRIAL: NCT02075294
Title: Efficacy and Safety Study of Adefovir and Entecavir for Elderly With Chronic Hepatitis B
Status: Completed | Type: Observational
Sponsor: Ying-Jie Ji (Other)
Responsible Party: Sponsor-Investigator, Ying-Jie Ji, MD, Beijing 302 Hospital
Organization: Beijing 302 Hospital (Other)
Other Study IDs: YNKT201313
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Hepatitis B, Chronic
Keywords: Aged; Hepatitis B, Chronic; Antiviral Agents
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — adefovir dipivoxil; entecavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- youth: <45years
  Adefovir dipivoxil or Entecavir
  Participants who received 10mg ADV more than 3 years or switch to other agent due to Renal dysfunction will be recruited.
  Participants who received 0.5mg ETV more than 3 years will be recruited.
  Interventions: Drug: Adefovir dipivoxil or Entecavir
- middle age: ≥45years and<65years
  Adefovir dipivoxil or Entecavir
  Participants who received 10mg ADV more than 3 years or switch to other agent due to Renal dysfunction will be recruited.
  Participants who received 0.5mg ETV more than 3 years will be recruited.
  Interventions: Drug: Adefovir dipivoxil or Entecavir
- elderly: ≥65 years
  Adefovir dipivoxil or Entecavir
  Participants who received 10mg ADV more than 3 years or switch to other agent due to Renal dysfunction will be recruited.
  Participants who received 0.5mg ETV more than 3 years will be recruited.
  Interventions: Drug: Adefovir dipivoxil or Entecavir

INTERVENTIONS:
Drug: Adefovir dipivoxil or Entecavir — Adefovir tablet, 10mg, take orally, once per day, more than 3years, exact duration depend on specific conditions and guidelines.
  Entecavir tablet, 0.5mg, take orally, once per day, more than 3years, exact duration depend on specific conditions and guidelines
  Other Names: ADV, Hepsera,; ETV, Baraclude

SUMMARY:
It is estimated that 350-400 million people have chronic infection with hepatitis B virus (HBV) all over the world. In china, 93 million individuals suffer from this chronic condition. Currently, seven medications are approved for the treatment of hepatitis B: two formulations of interferon and four nucleos(t)ide analogues. The Chinese population has one of the longer average life spans, and the size of the aged population has been increasing rapidly. As a result, the prevalence of elderly patients with HBV has increased, and the potential for development of cirrhosis or hepatocellular carcinoma in such patients is real. Hence, treatment of elderly patients with HBV is an important issue. However, ADV or ETV has become first choice due to the more side effect of INF and the resistant of LAM and LdT. But treatment outcomes with ADV and ETV in elderly are not known yet. In this study, we will evaluate and compare the efficacy and tolerability of ADV and ETV between younger and older patients with HBV. The aims of the present study are (1)to assess the benefits of ADV or ETV therapy for elderly patients with chronic hepatitis B, and (2)to determine differences in the emergence rate of side effect.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years
2. HBsAg positive for more than 6 months before enrollment
3. Serum HBVDNA >2×104IU/ml and serum ALT >80U/L or TBIL < 34 umol/L for chronic hepatitis B
4. Serum ALT < 80U/L, but hepatic inflammation scores ≥ G2 or hepatic fibrosis stage ≥ S2 for chronic hepatitis B
5. Serum HBVDNA >40 IU/ml for cirrhosis regardless of ALT and TBIL

Exclusion Criteria:

1. Co-infected with HCV, HDV or HIV, or autoimmune liver diseases combined
2. received antiviral therapy or immunosuppressant drugs before 6 months prior to enrollment
3. Renal function: creatinine >1.5 ULN or eGFR< 50ml/min/1.73m2 before therapy
4. Combined with hepatocarcinoma before therapy
5. suspend therapy voluntarily
6. use other nephrotoxic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We retrospectively analyzed a consecutive cohort of chronic hepatitis B patients treated with ADV, 10mg, daily, or with ETV，0.5mg，daily between January 2010 and December 2013 in a single tererral referral hospital in Beijing. Data were retrieved from a prospectively maintined database.
Sampling Method: Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2010-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
the rates of serum HBVDNA undetectable and Renal dysfunction | 3years

SECONDARY OUTCOMES:
the rate of normalisation of ALT | at week 2、4、12、24、36、48、60、72、84、96
the rate of HBsAg negative | at week48、96、144
the rate of HBeAg seroconversion | at week 24、48、72、96、120、144
the rate of HBeAg negative | at week 24、48、72、96、120、144

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Jie Ji, MD., Principal Investigator — Beijing 302 Hospital
Locations (1):
- 302 military hospital of China, Beijing, Beijing Municipality, China

REFERENCES:
- See also: Click here for more recruit information about this study — http://www.302hospital.com/Html/Index.html